CLINICAL TRIAL: NCT03298269
Title: Behavioral Interventions for Chronic Pain and Opioid-Related Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1618
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement (Experimental)
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement
- Supportive Counseling (Active Comparator)
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention led by a therapist that combines training in mindfulness, cognitive reappraisal, and savoring skills.
  Other Names: MORE
  Arms: Mindfulness-Oriented Recovery Enhancement
Behavioral: Supportive Counseling — A support group led by a therapist will allow participants to express emotions, share experiences, and receive social support.
  Other Names: Support Group
  Arms: Supportive Counseling

SUMMARY:
The purpose of this study is to examine the effects of Mindfulness-Oriented Recovery Enhancement versus a social support group (supportive counseling) intervention for chronic pain patients receiving long-term opioid pharmacotherapy for pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60+
* Current chronic pain condition
* Current use of prescription opioid agonist or mixed agonist-antagonist analgesics for >90 days

Exclusion Criteria:

* Prior experience with Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, or Mindfulness-Based Relapse Prevention
* Active suicidality, schizophrenia, psychotic disorder, and/or severe substance dependence (other than opioid dependence)
* Opioid misuse as determined by Current Opioid Misuse Measure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in pain symptoms | Change from baseline through study completion (9 months post-treatment)
  Pain severity and interference as measured by the Brief Pain Inventory
Change in aberrant drug-related behaviors | Change from baseline through study completion (9 months post-treatment)
  Aberrant drug-related behaviors as evidenced by triangulated aggregate of Current Opioid Misuse Measure and/or clinician assessment via Addiction Behaviors Checklist and/or urine screen

SECONDARY OUTCOMES:
Change in emotional distress | Change from baseline through study completion (9 months post-treatment)
  Distress measured by the Depression, Anxiety, Stress Scale
Change in opioid dose | Change from baseline through study completion (9 months post-treatment)
  Opioid dose converted into morphine equivalents via standardized equianalgesic tables
Change in opioid craving | Change from baseline through study completion (9 months post-treatment)
  Craving measured by visual analogue scale
Change in interoceptive awareness | Change from baseline through 8 weeks
  Interoceptive awareness measured by the Multidimensional Assessment of Interoceptive Awareness
Change in reappraisal | Change from baseline through 8 weeks
  Reappraisal measured by the Emotion Regulation Questionnaire
Change in savoring | Change from baseline through 8 weeks
  Savoring measured by the brief Ways of Savoring checklist
Change in meditative experiences | Change from baseline through 8 weeks
  As measured by the Five Facet Mindfulness Questionnaire, self-salience and self-extension items, and/or Nondual Awareness Dimensional Assessment
Change in body sensations | Change from baseline through 8 weeks
  Change in pleasant, neutral, and unpleasant body sensations as measured by body map

OTHER OUTCOMES:
Change in cue-reactivity | Change from baseline through 8 weeks
  Change in EEG responses during a cue-reactivity task
Change in emotion regulation | Change from baseline through 8 weeks
  Change in EEG responses during an emotion regulation task

CONTACTS AND LOCATIONS:
Locations (1):
- College of Social Work, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garland EL, Hudak J, Hanley AW, Nakamura Y. Mindfulness-oriented recovery enhancement reduces opioid dose in primary care by strengthening autonomic regulation during meditation. Am Psychol. 2020 Sep;75(6):840-852. doi: 10.1037/amp0000638. PMID 32915027
- [Derived] Garland EL, Hanley AW, Riquino MR, Reese SE, Baker AK, Salas K, Yack BP, Bedford CE, Bryan MA, Atchley R, Nakamura Y, Froeliger B, Howard MO. Mindfulness-oriented recovery enhancement reduces opioid misuse risk via analgesic and positive psychological mechanisms: A randomized controlled trial. J Consult Clin Psychol. 2019 Oct;87(10):927-940. doi: 10.1037/ccp0000390. PMID 31556669